CLINICAL TRIAL: NCT03896984
Title: DescriPtive Analysis of Real-world Clinical Outcomes of Second Line (2L) Novel Anti-HormonE Therapy (NAH) or RadIum-223 (Xofigo) in Patients With Metastatic Castration Resistance Prostate Cancer (mCRPC) After First Line (1L) NAH Therapy
Brief Title: Descriptive Analysis of Clinical Outcomes in Patients With Prostate Gland Cancer, Which Spreads to Other Parts of the Body, Who Were Treated First With Novel Anti-hormone Therapy Followed by a Second Line Treatment With Novel Anti-Hormone Therapy or RadIum-223 (Xofigo).
Acronym: PHENIX
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20526
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — Radium-223; radium Ra 223 dichloride; abiraterone; enzalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort_2LX: Patients with mCRPC who received NAH monotherapy (Abiraterone or Enzalutamide) as first liine (1L) after diagnosis of mCRPC who then received Ra-223 monotherapy as second line (2L) treatment
  Interventions: Drug: Radium-223 (Xofigo, BAY88-8223); Drug: Abiraterone; Drug: Enzalutamide
- Cohort_2LH: Patients with mCRPC who received NAH monotherapy (Abiraterone or Enzalutamide) as 1L after diagnosis of mCRPC who then received another NAH monotherapy (i.e., Abiraterone to Enzalutamide or Enzalutamide to Abiraterone) as 2L treatment. None of the patients had ever received Radium-223 dichloride
  Interventions: Drug: Abiraterone; Drug: Enzalutamide

INTERVENTIONS:
Drug: Radium-223 (Xofigo, BAY88-8223) — Ra-223 was approved by the FDA in May 2013 for the treatment of patients with castration-resistant prostate cancer, symptomatic bone metastases and no known visceral metastatic disease.
  Groups: Cohort_2LX
Drug: Abiraterone — Abiraterone is a CYP17 inhibitor. It was approved by the FDA for the treatment of patients with mCRPC in 2011, and for patients with metastatic high-risk castration-sensitive prostate cancer in 2018.
Drug: Enzalutamide — Enzalutamide is an androgen receptor inhibitor. It was approved by the FDA for the treatment of patients with mCRPC in 2012, with warning and precautions added in 2017 regarding the risk of seizure and encephalopathy.

SUMMARY:
In this study researcher want to learn more about the overall survival in patients suffering from prostate gland cancer which spread outside the prostate to other parts of the body who received either a novel anti-hormone therapy (NAH) or Radium-223 (Xofigo) after a prior NAH therapy (first line treatment). Additionally the researchers are also interested in the occurrence of bone fractures and other skeletal events. Basis for this study will be the US based Flatiron database which provides access to clinical data for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented mCRPC receiving 1L NAHs.
* Initiation of Ra-223 after 1L NAH therapy, or
* Initiation of sequential NAH therapy after 1L NAH therapy

Exclusion criteria:

* Patients involved in clinical trials
* Patients who received combined therapies in 1L or 2L

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The primary study population consists of patients with documented mCRPC who either received Ra-223 or sequential NAH therapy after 1L NAH therapy respectively.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) from initiation of 2L therapy of Radium-223 in patients with mCRPC after 1L NAH therapy | Retrospective analysis from 2013-01-01 to 2018-12-30
Overall survival (OS) from initiation of 2L therapy of sequential NAH in patients with mCRPC after 1L NAH therapy | Retrospective analysis from 2013-01-01 to 2018-12-30

SECONDARY OUTCOMES:
Descriptive analysis of patient demography at baseline | Retrospective analysis from 2013-01-01 to 2018-12-30
  Demographic characteristics includes:
  * Gender (expecting 100% male)
  * Age (in the year of index date)
  * Ethnicity
Descriptive analysis of clinical characteristics of patients at baseline | Retrospective analysis from 2013-01-01 to 2018-12-30
  Clinical characteristics includes:
  * Histology
  * Gleason score
  * Clinical stage (at initial diagnosis)
  * T/N/M stage (at initial diagnosis)
  * ECOG performance status
  * Site of metastasis (visceral, lymph node, bone)
Descriptive analysis of laboratory values at baseline | Retrospective analysis from 2013-01-01 to 2018-12-30
  The laboratory tests of interest includes:
  * Prostate Specific Antigen(PSA)
  * Alkaline Phosphatase(ALP)
  * Hemoglobin (Hgb)
  * Lactate dehydrogenase (LDH)
Frequency of SSEs of Radium-223 versus Abiraterone or Enzalutamide after 2L | Retrospective analysis from 2013-01-01 to 2018-12-30
  SSE:Symptomatic skeletal event
Incidence rate of SSEs of Radium-223 versus Abiraterone or Enzalutamide after 2L | Retrospective analysis from 2013-01-01 to 2018-12-30
Frequency of pathologic fracture of Radium-223 versus Abiraterone or Enzalutamide after 2L | Retrospective analysis from 2013-01-01 to 2018-12-30
Incidence rate of pathologic fracture of Radium-223 versus Abiraterone or Enzalutamide after 2L | Retrospective analysis from 2013-01-01 to 2018-12-30
Period of time from initiation of 2L to first SSE | Retrospective analysis from 2013-01-01 to 2018-12-30

CONTACTS AND LOCATIONS:
Locations (1):
- US Flatiron prostate cancer database, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Result] Sartor O, George D, Tombal B, Agarwal N, Higano CS, Sternberg CN, Miller K, Jiao X, Guo H, Sandstrom P, Bruno A, Verholen F, Saad F, Shore N. Real-world outcomes of second novel hormonal therapy or radium-223 following first novel hormonal therapy for mCRPC. Future Oncol. 2022 Jan;18(1):35-45. doi: 10.2217/fon-2021-0886. Epub 2021 Oct 12. PMID 34636627